CLINICAL TRIAL: NCT05570682
Title: Manually Controlled Infusion Vs Target Controlled Infusion: an Hemodynamic Alterations in StrokeThrombectomy Evaluation (HASTE); a Multi-center Randomized Controlled Trial
Brief Title: Manually Controlled Infusion Vs Target Controlled Infusion for StrokeThrombectomy
Acronym: HASTE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No particpants was enrolled as after IRB cleareance there was no more logistical feasibiliy to enroll patients.
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Alessandro De Cassai, Medical Doctor, University of Padova
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HASTE
Record Dates: First submitted 2022-09-30; First posted 2022-10-06 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Stroke, Ischemic; Stroke/Brain Attack; Anesthesia; Hemodynamic Instability
MeSH Terms: conditions — Ischemic Stroke; Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants undergoing intervention will be unaware of the intervetion Outcomes assessor will be not involted in the other study of the study and will be not aware of the intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Manual induction (Active Comparator): General Anesthesia induction: Fentanyl 2 mcg/kg, Propofol 2 mg/kg, Rocuronium 0.6 mg/kg General Anesthesia mainteneance: Propofol 4-6 mg/kg/h to keep an adequate sedation level (BIS between 40-60; entropy between 40-60)
  Interventions: Procedure: Manual induction
- Target Controlled Induction (Experimental): General Anesthesia induction: Fentanyl 2 mcg/kg, Propofol TCI with Schneider site effect model starting from 2 mcg/ml and increasing the dose untile loss of consciousness, Rocuronium 0.6 mg/kg.
  General Anesthesia mainteneance: Propofol TCI with Schneider site effect model in order to keep an adequate sedation level (BIS between 40-60; entropy between 40-60)
  Interventions: Procedure: TCI

INTERVENTIONS:
Procedure: TCI — General anesthesia will be induced with a TCI pump
  Arms: Target Controlled Induction
Procedure: Manual induction — General anestehsia will be induced and maintained using a pro kilo regimen.
  Arms: Manual induction

SUMMARY:
The goal of this randomized controlled trial is to compare manual general anesthesia induction to general anesthesia induction guided by target controlled infusion system in cerebral ischemic stroke

The main questions it aims to answer are:

* Does target controlled infusion has a more favorauble hemodynamic profile than manual general anesthesia induction?
* Do patients receiving general anesthesia with target controlled infusion system have a more favourable outcome? Participants will receive general anesthesia induction with a target controlled infusion system and will be compared to patients receiving manual general anesthesia induction.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Anterior Cerebral Circulation Stroke
* Patient eligible for mechanical trombectomy
* mRS ≤ 2;
* Fasting patients (>6 h solid, >2 hours liquids)
* Glashow Coma Scale more than seven.

Exclusion criteria

* Patient in general anesthesia at hospital arrival
* Associated hemorrhagic stroke

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-10-09 (Actual); Primary Completion 2022-10-09 (Actual); Study Completion 2022-10-09 (Actual)

PRIMARY OUTCOMES:
Number of patients with Intraprocedural Hypotension | Up to three hours
  Descrease of mean blood pressure > 20% during the procedure from the baseline

SECONDARY OUTCOMES:
Change from baseline in National Institutes of Health Stroke Scale at 24 hours after acute ischemic stroke | 24 hours after acute ischemic stroke
  Change from baseline in National Institutes of Health Stroke Scale (NIHSS) at 24 hours after acute ischemic stroke. The NIHSS is composed of 11 items, each of which scores a specific ability between a 0 and 4. For each item, a score of 0 typically indicates normal function in that specific ability, while a higher score is indicative of some level of impairment.The individual scores from each item are summed in order to calculate a patient's total NIHSS score. The maximum possible score is 42, with the minimum score being a 0
Change from baseline in National Institutes of Health Stroke Scale at 7 days after acute ischemic stroke | 7 days after acute ischemic stroke
  Change from baseline in National Institutes of Health Stroke Scale (NIHSS) at 7 days after acute ischemic stroke. The NIHSS is composed of 11 items, each of which scores a specific ability between a 0 and 4. For each item, a score of 0 typically indicates normal function in that specific ability, while a higher score is indicative of some level of impairment.The individual scores from each item are summed in order to calculate a patient's total NIHSS score. The maximum possible score is 42, with the minimum score being a 0
Evaluation of Modified Rankin Scale at 3 months after acute ischemic stroke | 3 months after acute ischemic stroke
  Evaluation of Modified Rankin Scale at 3 months after acute ischemic stroke. Modified Rankin Score is a 6 point disability scale with possible scores ranging from 0 to 5. A separate category of 6 is added for patients who expire.
Percentage of patients alive at 3 months after acute ischemic stroke | 3 months after acute ischemic stroke
  Percentage of patients alive at 3 months after acute ischemic stroke
Difference in modified treatment in cerebral infarction (mTICI) score | 24 hours after ischemic stroke
  Successfull reperfusion in the two groups will be evaluated by modified tratment in cerebral infarction score. modified treatment in cerebral infarction is a five point score (0,1,2a,2b,3) with 0 menaning o reperfusion and 3 complete reperfusion
Difference in time from door to groin | Up to 6 hours
  Time will be evaluated from patient admission to the beginning of angiographic procedure
Difference in time from groin to reperfusion | Up to 6 hours
  It will be evaluated the overall time of angiographic procedure
Difference in Intensive Care Unit/Stroke Unit stay | Up to 30 days
  Overall patient stay in intensive care unit/stroke unit in days

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Padova, Padua, Veneto, Italy